CLINICAL TRIAL: NCT03549780
Title: A Pilot Study of a Novel Stomal Occlusion Device in Patients With a Brooke Ileostomy
Brief Title: Novel Stomal Occlusion Device in Patients With a Brooke Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William A. Faubion, M.D. (Other)
Responsible Party: Sponsor-Investigator, William A. Faubion, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-001427
Record Dates: First submitted 2018-05-16; First posted 2018-06-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Ileostomy - Stoma
Keywords: Brooke Ileostomy; stoma; ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Stomal Occlusion (Other): Insertion of a novel stomal occlusion device into patients with Brooke Ileostomy and assess feasibility and patient satisfaction
  Interventions: Device: Stomal Occlusion Device

INTERVENTIONS:
Device: Stomal Occlusion Device — Insertion of a novel stomal occlusion device into patients with Brooke Ileostomy and assess feasibility and patient satisfaction

SUMMARY:
This investigation constitutes an initial evaluation of the stoma occlusion device in humans with a mature permanent Brooke ileostomy. The overall objective of this study is to assess feasibility and initial operating characteristics of a novel stoma occlusion device. The study will recruit 20 patients for placement of the device into the mature Brooke ileostomy and subsequent 2 hour observation period. The device will remain in the ileostomy for up to 2 hours.

DETAILED DESCRIPTION:
An ostomy is a protrusion of part of the intestines extending through the abdominal wall for the purpose of elimination of wastes and may be temporary or permanent depending on the purpose of the initial surgery. The most common reasons for permanent bowel diversion are cancer and ulcerative colitis. Appliances have improved greatly over the last 50 years, but patients continue to experience appliance leakage and skin infections and struggle with the emotional and social impact of an external pouch. This study seeks to answer the opportunity to significantly improve quality of life to a large segment of the global population through optimization of a technology for a stoma occlusion device in patients with permanent stomas. Four pre-clinical animal studies have been conducted. All the animals that completed the study tolerated the device well and had no adverse reactions to device materials. This project will allow a prototype of an artificial stomal occlusion device to be tested in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 and older
* Gender: Male and Female
* Target disease or condition: 20 patients with permanent End Ileostomy, specifically Brooke ileostomy for greater than 3 years
* Ability to comply with protocol
* Competent and able to provide written informed consent

Exclusion Criteria:

* Inability to provide consent
* Crohn's Disease
* Koch pouch
* Pregnancy
* If subject's stoma length is less than 4 cm or longer than 8 cm
* Clinically significant medical conditions within the six months before participation with the device that would, in the opinion of the investigators, compromise the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 hours
  Safety: Device is able to be inserted adequately (function) and without any significant patient discomfort or adverse events (safety).

SECONDARY OUTCOMES:
Function (continence of device); observed leakage | 2 hours
  Device is able to be inserted adequately (function) and without any significant patient discomfort or adverse events (safety). The function (continence) of the stoma occlusion device: After the device has been inserted, a 4 x 4 inch gauze will be placed at the stoma site and secured in place. The gauze functions to document any moisture or leakage of the occlusion device. Consistency and volume of moisture or leakage on the gauze pad will be documented.

OTHER OUTCOMES:
Questionnaire | 2 hours
  The patients' overall satisfaction/acceptance with the device: Patient satisfaction/acceptance will be documented on a questionnaire that will be administered to them after the study visit is completed. 10 questions, Likert scale design.

CONTACTS AND LOCATIONS:
Overall Officials: William A Faubion, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials